CLINICAL TRIAL: NCT01388699
Title: Migraine and Endothelial Dysfunction
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Thomas Liman, MD MSC, Charite University, Berlin, Germany
Other Study IDs: FF_NCRC_Migraine&ED
Record Dates: First submitted 2011-07-05; First posted 2011-07-07 (Estimated); Last update posted 2018-07-18 (Actual); Status verified 2018-07

CONDITIONS: Migraine With Aura
Keywords: Migraine with aura
MeSH Terms: conditions — Migraine with Aura

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- migraine group: female migraineurs with aura
- control group: healthy women without headache syndrome

SUMMARY:
Recently, there is evidence that endothelial activation and dysfunction are associated with migraine, especially in female migraineurs with aura. Our objectives were to determine whether novel endothelial function markers are altered in female migraineurs with aura compared to age-matched controls.

DETAILED DESCRIPTION:
Our objectives were to determine whether novel endothelial function methods and novel markers of endothelial activation are associated with migraine in female migraineurs with aura.

Migraine is an independent risk factor for stroke, especially in young women with aura symptoms. Endothelial dysfunction is a risk factor for cardiovascular diseases. Recent studies suggest that there is a link between migraine with aura and endothelial activation, dysfunction and impaired vascular reactivity.

In this case-control study the investigators examine several novel biomarkers of endothelial function such as endothelial progenitor cells and endothelial microparticles as well as novel methods such as reactive hyperemic peripheral arterial tonometry in female migraineurs with aura and age-matched controls.

ELIGIBILITY:
Inclusion Criteria:

* migraine with aura
* age < 50
* female gender

Exclusion Criteria:

* severe infectious disease
* cardiovascular disease (stroke, coronary heart disease, myocardial infarction)
* vasculitis
* peripheral artery disease
* diabetes mellitus
* pregnancy
* drug abuse
* medication: statin, anticoagulation, aspirin, clopidogrel
* intake of triptans <24h

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: female migraineurs from outpatient clinic
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2010-10; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Endothelial Microparticles | baseline
  Levels of endothelial microparticlel in the peripheral blood using flow cytometry

SECONDARY OUTCOMES:
Levels of circulating Endothelial Progenitor Cells | baseline
  Levels of cEPC (CD34+/CD133+/VGF2R/CD31) in % of mononuclear cells using flow cytometry
Digital pulse volume change | baseline
  Digital pulse volume change (with RH PAT as non invasive measurement (PAT-ratio; ENDOPAT, Itamar Medical Ltd.) for non-invasive, peripheral endothelial function

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Liman, MD, Principal Investigator — Center for Stroke Research Berlin, Charité Campus Mitte
Locations (1):
- Center for Stroke Research Berlin, Berlin, Germany

REFERENCES:
- [Background] Liman TG, Neeb L, Rosinski J, Wellwood I, Reuter U, Doehner W, Heuschmann PU, Endres M. Peripheral endothelial function and arterial stiffness in women with migraine with aura: a case-control study. Cephalalgia. 2012 Apr;32(6):459-66. doi: 10.1177/0333102412444014. Epub 2012 Apr 20. PMID 22523187
- [Background] Liman TG, Bachelier-Walenta K, Neeb L, Rosinski J, Reuter U, Bohm M, Endres M. Circulating endothelial microparticles in female migraineurs with aura. Cephalalgia. 2015 Feb;35(2):88-94. doi: 10.1177/0333102414529671. Epub 2014 Apr 8. PMID 24715500
- [Background] Liman TG, Neeb L, Rosinski J, Reuter U, Endres M. Stromal Cell-Derived Factor-1 Alpha Is Decreased in Women With Migraine With Aura. Headache. 2016 Sep;56(8):1274-9. doi: 10.1111/head.12839. Epub 2016 May 30. PMID 27238143